CLINICAL TRIAL: NCT03897400
Title: Evaluation of Ovarian Reserve in Crohn's Disease
Brief Title: Ovarian Reserve in Crohn's Disease
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pınar Kadirogulları, pınar kadiroğulları, M.D, Department of Obstetrics and Gynecology, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: 2019.03.40
Record Dates: First submitted 2019-03-27; First posted 2019-04-01 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Crohn Disease; Ovary Disease; Anti-Mullerian Hormone Deficiency
MeSH Terms: conditions — Crohn Disease; Ovarian Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group: women in reproductive age with crohn's disease
  Interventions: Other: AMH levels in young women with crohn's disease will be considered.
- control group: women in reproductive age without crohn's disease,
  Interventions: Other: AMH levels in young women with crohn's disease will be considered.

INTERVENTIONS:
Other: AMH levels in young women with crohn's disease will be considered. — Ovarian Reserve in Young Women of Reproductive Age with Crohn's Disease;Blood will be taken from both the study and control groups and the AMH level will be evaluated.

SUMMARY:
Crohn's disease reduces fertility by inducing inflammation both directly and in the fallopian tubes and ovaries and indirectly through surgical interventions and tubal adhesions associated with disease treatment. Anti-mullerian hormone (AMH) is a reliable indicator of ovarian reserve in women. The aim of this study was to compare serum AMH levels in women with Crohn's disease and healthy controls. In this study, the investigators aimed to investigate AMH and ovarian capacity in the study group with crohn's disease and in the control group without disease.

ELIGIBILITY:
Inclusion Criteria:

* crohn's disease;
* reproductive age women

Exclusion Criteria:

* Over 40 years old,
* a previous ovarian resection;
* renal failure (serum creatinine levels N1.2 mg / dL);suspicion of malignancy;
* the presence of hereditary or acquired hematological disease;
* pregnancy;
* current lactation;
* the presence of a serious comorbid chronic disease;
* cirrhosis originating from chronic liver disease;
* abnormal thyroid function tests;
* a known serious psychological problem;
* presence of alcoholism and male sex.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study group consisted of young women in the reproductive age with crohn's disease.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
AMH levels | 1 MONTH
  AMH levels of subjects taken into groups will be evaluated in lg/L

SECONDARY OUTCOMES:
ultrasound findings | 1 MONTH
  On the 3rd day of the menstrual cycle, the patients will be given ultrasound and the ovarian volume will be examined. the ovarian volume will be calculated by taking the size of the ovary in three sections.

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Süleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)